CLINICAL TRIAL: NCT02179177
Title: Impact of Daily Prophylaxis Dose Anticoagulation With a Factor Xa Inhibitor (Apixaban) in Patients With Sickle Cell Disease
Brief Title: Apixaban in Patients With Sickle Cell Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: funding has been exhausted
Sponsor: Nirmish Shah (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Nirmish Shah, Assistant Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00048953
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Vaso-occlusive Crisis; Reduction in Hospitalizations; Sickle Cell Disease
Keywords: Vaso-occlusive crisis; Reduction in hospitalizations; Sickle Cell Disease
MeSH Terms: conditions — Vaso-Occlusive Crises; Anemia, Sickle Cell | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Active Comparator): Active drug Apixaban 2.5mg taken by mouth twice a day
  Interventions: Drug: Apixaban
- Placebo (Placebo Comparator): Sugar pills that look like Apixaban that will be taken by mouth twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apixaban — Drug is taken by mouth twice a day for 6 months
  Arms: Apixaban
Drug: Placebo
  Arms: Placebo

SUMMARY:
In patients with SCD, the use of low dose anticoagulation as an outpatient may lead to a significant decrease in morbidity and as a result, decrease healthcare utilization and costs. This study attempts to critically avoid admissions by reducing daily pain scores and pain crisis as an outpatient by use of a novel oral anticoagulant.

DETAILED DESCRIPTION:
There is not only significant morbidity associated with patients with SCD, but also costs associated with the numerous hospitalizations. Small studies have been unable to show clear benefit of the use of low dose anticoagulation in SCD due to limited sample size or the inclusion of very specific populations. However, studies have shown a decrease in the level of elevated prothrombotic markers with anticoagulation, and one study using full dose anticoagulation in patients with a generally milder form of SCD (with high protective hemoglobin) showed more rapid decrease in clinical pain with use of anticoagulation, suggesting a possible benefit of such therapy. Due to the paucity of data to support therapeutic dose LMWH in the more severe forms of SCD seen in the United States, we have chosen prophylactic dose anticoagulation. This study proposal attempts to critically avoid admissions by reducing daily pain scores and pain crisis as an outpatient by use of a novel oral anticoagulant.

The development of novel anticoagulants such as oral direct factor Xa (FXa) inhibitors allows the realistic use of daily prophylactic dosing as an outpatient. Past studies as detailed earlier have been limited by attempts to use subcutaneous injections or frequent, close monitoring for acenocoumarol treatment, both which are not ideal for chronic daily use. Furthermore, the use of global assays such calibrated automated thrombography (CAT) have shown further details about thrombin generation in a population which is hypercoagulable at baseline.

This is a double blind, parallel group, placebo controlled feasibility study with an enrollment target of 25 patients (12 per arm). All subjects that meet inclusion criteria as an outpatient, following a 1 month observation, will be randomized to receive an oral prophylactic dose factor Xa inhibitor (Apixaban 2.5mg po bid) or placebo for 6 months. Subjects will return for a 30 day (+/- 5 days) follow-up visit after the End of Treatment (EOT) visit. Initial randomization will occur by computerized randomization technique by the investigational drug services (IDS) at Duke University Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* documented HgbSS, SC or HgbS-beta0 thalassemia,
* age ≥18 years old and ≤80,
* seen in outpatient clinic ≥2 times in past year
* seen for an acute care visit (hospitalization, emergency department, or day hospital visit) for pain >2 times in the past year.

Exclusion Criteria:

* Hospitalization or day hospital visit for pain crisis within the past 2 weeks
* Patients with ≥10 acute care visits within the past year will be excluded
* Creatinine >3.0 mg/dL
* creatinine ≥1.5 mg/dL AND weight ≤60 kg
* chronic use of antiplatelet or anticoagulation medication
* Patients with known vasculopathy or Moya-Moya
* platelet count <100 X 109/L
* AST or ALT >3 times normal
* chronic red blood cell transfusions (scheduled transfusions)
* packed red blood cell transfusion within the past 2 months
* Use of CYP3A4 and P-gp inhibitor medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2017-09-03 (Actual); Study Completion 2017-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirmish Shah, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with sickle cell disease were enrolled as an outpatient in clinic while at baseline pain from January 2015 to September 2017.
Groups:
- Placebo: Sugar pills that look like Apixaban that will be taken by mouth twice a day
  Placebo
Period: Overall Study
Arm/Group | Apixaban | Placebo
Started | 8 | 8
Completed | 6 | 6
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (6.2) | 33 (3.9) | 31.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain as Measured by Visual Analog Scale (VAS)
Description: The primary pain assessment tool will be a 10-cm horizontal visual analog scale (VAS), with "0" corresponding to no pain at one end and "10" indicating the worst pain at the other.
Time Frame: Month 1 to Month 8
Population: Two participants in each group (Apixaban and Placebo) did not return for Month 8 visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apixaban | Placebo
Number analyzed (Participants) | 6 | 6
score on a scale | -1 (0.5) | 0 (0.4)
Statistical Analysis 1: Comparison: Apixaban vs Placebo; Test type: Other; p = 0.11, t-test, 2 sided; Mean Difference (Net) = 1

2. Secondary Outcome: Change in Thrombin Generation Using D-dimer Measurement as a Surrogate
Time Frame: Enrollment to 2 months
Population: Data not collected.
Arm/Group | Apixaban | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Daily Pain Scores While Hospitalized as Measured by VAS
Description: The primary pain assessment tool will be a 10-cm horizontal visual analog scale (VAS), with "0" corresponding to no pain at one end and "10" indicating the worst pain at the other. Secondary analysis will be performed to evaluate differences when patients are hospitalized and on study drug versus placebo.
Time Frame: up to 8 months
Population: Two participants from each group (Apixaban and Placebo) did not return for Month 8 visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apixaban | Placebo
Number analyzed (Participants) | 6 | 6
score on a scale | 6.4 (3.4) | 6.6 (3.8)

4. Secondary Outcome: Number of Hospitalizations During Treatment
Time Frame: up to 8 months
Population: Two participants from each group (Apixaban and Placebo) did not return for 8 Month visit.
Measure: Mean (Standard Deviation); unit: hospitalizations
Arm/Group | Apixaban | Placebo
Number analyzed (Participants) | 6 | 6
hospitalizations | 3 (3.3) | 1.5 (1.5)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Apixaban | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=8) | Placebo (N=8)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Hospitalization (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=8) | Placebo (N=8)
Sickle Cell Crisis (Cardiac disorders) | 1 | 0
Sickle Cell Crisis (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT02179177/Prot_SAP_000.pdf